CLINICAL TRIAL: NCT05229159
Title: Bio Impedance Electrical Analysis to Predict Outcome After Cardiac Surgery
Acronym: BiPOCS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 456
Record Dates: First submitted 2021-11-22; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Care After Cardiac Surgery With Cardio Pulmonary Bypass
Keywords: phase angle; cardiac surgery; cardiopulmonary bypass; risk stratification; outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BiPOCS group: All patients of our centers admitted for postoperative care after cardiac surgery with cardiopulmonary bypass and receiving a bioelectrical impedance analysis at the admission.
  Interventions: Diagnostic Test: Bioelectrical impedance analysis

INTERVENTIONS:
Diagnostic Test: Bioelectrical impedance analysis — Segmental multi-frequency bioelectrical impedance analysis are carried out at all patient admitted to our ICU for postoperative care after cardiac surgery with cardiopulmonary bypass. Our objective is to evaluate the relevance of phase angle to predict mortality or a prolonged hospital length of stay. Phase angle is evaluated at ICU admission and will be compared to well-known prognostic scores computed in preoperative (EuroSCORE II) and at day one after surgery (SOFA, CASUS and SAPS II).

SUMMARY:
Phase angle determined by bioelectrical impedance analysis is a strong prognostic factor in several medical areas as clinical nutrition, nephrology, infectious disease, oncology. Inflammation, frailty status and fluid overload can lead to a phase angle decreased. Some studies support its use for risk stratification in intensive care unit and other in preoperative for cardiac surgery. The investigators would like to evaluate its relevance for risk stratification at intensive care unit admission in the context of postoperative cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18
* Cardiac surgery with cardiopulmonary bypass
* Bioelectrical impedance analysis the day of the admission in intensive care unit

Exclusion Criteria:

* Left ventricular assist device
* Limitations des thérapeutiques actives en place pour le patient
* Patient opposition to the use of his health data
* Invalid bioelectrical impedance analysis
* Advanced directives to withhold or withdraw life-sustaining treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients admitted in intensive care unit for postoperative care after cardiac surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve to predict a composite criterion including in-hospital mortality or prolonged hospital length of stay. | at 6 months after the cardiac surgery
  The phase angle's area under the receptor operative curve to predict a composite criteria evaluated at hospital discharge and combining:
  * In hospital mortality
  * Prolonged hospital length of stay, defined by an in hospital length of stay greater than the 75th percentile of length of stay in the study population"

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital cardiologique Louis Pradel Groupe Hospitalier Est, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No